CLINICAL TRIAL: NCT06817447
Title: Prophylactic Pulmonary Vein Isolation in Typical Atrial Flutter and Heart Failure: a Prospective, Multi-center, Randomized Controlled Study
Brief Title: Pulmonary Vein Isolation in Typical Atrial Flutter and Heart Failure
Acronym: PVI-AFL-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Dr., The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-SR-026
Record Dates: First submitted 2025-01-25; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atrial Flutter Typical; Heart Failure
Keywords: atrial flutter; Heart failure; Pulmonary vein isolation
MeSH Terms: conditions — Heart Failure; Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Follow-up physicians are blinded to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTI-alone arm (Active Comparator)
  Interventions: Procedure: Cavo-tricuspid isthmus ablation
- CTI+CPVI Arm (Experimental)
  Interventions: Procedure: Pulmonary vein isolation plus cavo-tricuspid isthmus ablation

INTERVENTIONS:
Procedure: Pulmonary vein isolation plus cavo-tricuspid isthmus ablation — For those who are randomized to CTI+CPVI Arm, additional CPVI should be performed after finishing CTI ablation. CPVI could be performed using open-irrigated contact-force catheter, cryoballoon catheter or pulse-field ablation catheter. The endpoint is defined as both entrance and exit block in the pulmonary veins.
  Arms: CTI+CPVI Arm
Procedure: Cavo-tricuspid isthmus ablation — In periprocedural period, all antiarrhythmic drugs were discontinued for at least 5 half-lives and amiodarone for 2 months before the procedure. An electrophysiological study was performed after overnight fasting and mild sedated state with administration of intravenous midazolam and fentanyl.
  CTI ablation should be performed under the CARTO or Ensite electroanatomic mapping system using an open-irrigated contact-force ablation catheter. Radiofrequency should be delivered at 30-50 W with a contact-force between 5-30 g in a point-by-point fashion until the CTI line is completed. Touch-up radiofrequency should be performed as needed. The endpoint of ablation is termination of AFL, if present, and the demonstration of bidirectional block across the CTI by using differential pacing.
  Arms: CTI-alone arm

SUMMARY:
This study, called the PVI-AFL-HF Trial, investigates two treatments for patients with typical atrial flutter (AFL) and heart failure (HF). It aims to determine whether adding prophylactic pulmonary vein isolation (CPVI) to the standard cavo-tricuspid isthmus (CTI) ablation improves long-term outcomes compared to CTI ablation alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Typical AFL referring for ablation
* No prior history of AF
* Fulfilling the criteria for HF: New York Heart Association (NYHA) function class II or greater; and N-terminal pro-brain natriuretic peptide (NT-pro-BNP) >125 pg/ml in sinus rhythm or >365 pg/ml in AFL
* Optimized guideline-directed medical therapy for HF for at least one month
* A minimum of anticoagulation for three weeks
* Sign informed consent

Exclusion Criteria:

* Any AF episodes documented during 48-hour Holter monitoring
* Presence of left atrial thrombus
* HF due to infiltrative cardiomyopathy, constrictive pericarditis, active myocarditis, cardiac tamponade, or uncorrected primary valvular disease
* Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within three months prior to enrollment
* Previous cardiac transplantation, complex congenital heart disease, rheumatic heart disease
* Untreated hypothyroidism or hyperthyroidism
* Dialysis-dependent terminal renal failure
* Life expectancy <12 months due to non-cardiovascular causes.
* Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study
* Female under pregnancy or breast-feeding
* Involved in other studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of worsening heart failure requiring unplanned hospitalizations or urgent visits, and cardiovascular death | From randomization until completion of the planned follow-up, assessed up to 48 months

SECONDARY OUTCOMES:
Time to cardiovascular death | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to hospitalization or urgent visits for heart failure | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to hospitalization for heart failure | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to urgent visits for heart failure | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to all-cause death | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to atrial fibrillation recurrence | From randomization until completion of the planned follow-up, assessed up to 48 months
Time to change of diuretics | From randomization until completion of the planned follow-up, assessed up to 48 months
Change in quality of life - Kansas City Cardiomyopathy Questionnaire score (KCCQ-23) at one-year | One-year
  KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ Total Symptom Score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in 6-minute walk test at one-year | One-year
Change in N-terminal pro-B type natriuretic peptide (NT-proBNP) at one-year | One-year
Change in New York Heart Association (NYHA) class at one-year | One-year
  NYHA class is a widely used system for assessing the functional status and severity of heart failure symptoms in patients, with NYHA class IV being the worst.

IPD SHARING:
Plan to Share IPD: Undecided